CLINICAL TRIAL: NCT02393742
Title: Efficacy of Oral Sodium Nitrite for Improving Physiological Functions in Older Adults
Brief Title: Nitrite Supplementation for Improving Physiological Function in Older Adults
Acronym: NITRITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Douglas Seals, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: R01AG013038-19 (NIH)
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Ageing
MeSH Terms: interventions — Sodium Nitrite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Nitrite Supplementation (Experimental): 80 mg/day (40 mg 2x/day) slow release sodium nitrite (TheraVasc, Inc) for 3 months
  Interventions: Drug: Sodium nitrite
- Placebo (Placebo Comparator): placebo 2x/day for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium nitrite
  Arms: Sodium Nitrite Supplementation
Drug: Placebo
  Arms: Placebo

SUMMARY:
Nitric oxide (NO) is an essential molecule in the body that decreases with aging and causes reductions in vascular, movement ("motor") and cognitive functions. This study will determine if daily oral supplementation (3 months) with a compound that increases NO in the body, i.e., sodium nitrite, improves vascular, motor and cognitive function in older adults. The project also seeks to provide insight into the biological reasons (mechanisms) by which supplementation with sodium nitrite improves physiological function in older adults. Overall, this research will provide scientific evidence supporting the use of sodium nitrite for preserving physiological function and preventing clinical disease and disability with aging.

ELIGIBILITY:
Inclusion Criteria:

* • Age 60-79 years. Women will be confirmed as postmenopausal (either natural or surgical) based on cessation of menses for >1 year.

  * Ability to provide informed consent
  * Score >22 on the mini mental state exam (MMSE) to allow a broad range of normal and mildly-impaired cognitive abilities, but function adequate to understand and complete trials (214)
  * Baseline brachial flow-mediated dilation (FMD) < 7%Δ (rationale: non-invasive screening to ensure exclusion of subjects with exceptionally high baseline endothelial function(215))
  * Blood pressure (BP) >100/60 mmHg for past 3 mo (rationale: blood pressure below 100/60 mmHg may elevate the normally small risk of hypotension with sodium nitrite treatment)
  * Ability to perform motor and cognitive tests (e.g., can rise from a chair, walk for 2 min, climb 10 stairs)
  * Willing to accept random assignment to condition (older adults)

Exclusion Criteria:

* • High dietary nitrate intake or current nitrite supplementation; hypersensitivity to nitrates or nitrites

  * Glucose-6-phosphate dehydrogenase deficiency or blood methemoglobin >2%
  * Current smoking
  * Having past or present alcohol dependence or abuse, as defined by the American Psychiatry Association, Diagnostic and Statistical Manual of Mental Disorders
  * Body mass index (BMI) >40 kg/m2 (FMD measurements can be inaccurate in severely obese patients)
  * Chronic clinical diseases (e.g., coronary artery/peripheral artery/cerebrovascular diseases, diabetes, chronic kidney disease requiring dialysis, neurological disorders or diseases that may affect motor/cognitive functions [multiple sclerosis, Parkinson's disease, polio, Alzheimer's disease, dementia or other brain diseases of aging]), except hypertension and hyperlipidemia.
  * Regular vigorous aerobic/endurance exercise (>3 vigorous bouts/week)
  * Not weight stable in the prior 3 months (>2 kg weight change) or unwilling to remain weight stable throughout study (rationale: recent weight change or weight loss can influence vascular function and small metabolite signature(216))
  * Current treatment or recent cessation (< 3 mo) of hormone replacement therapy.
  * Moderate or severe peripheral artery disease (ankle-brachial index <0.7)(183)
  * A graded exercise test will be performed by all subjects, if there is physician concern or an adverse event, the subject will not participate in a maximal oxygen consumption test (this will be determined in accordance with stated contraindications for exercise testing provided by the American Heart Association)(217)
  * Claustrophobia, metal implants, etc., affecting feasibility and/or safety of the fMRI scanning.

Ages: 60 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Vascular Function | 3 months
  flow mediated dilation
Motor Function | 3 months
  rate of torque development

SECONDARY OUTCOMES:
Systemic oxidative stress and inflammation | 3 months
  circulating markers of oxidative stress and inflammation
Number of participants with additional measures of motor ability | 3 months
  tests of balance, endurance, strength, and dexterity
endothelial cell oxidative stress and inflammation | 3 months
  inflammatory and oxidative stress markers in biopsied endothelial cells
plasma metabolites | 3 months
NIH Toolbox cognition test battery | 3 months
  Cognitive Function

OTHER OUTCOMES:
neural activation | 3 months
  brain activity measured during n-back task in functional magnetic resonance imaging (fMRI)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Rossman, PhD, Study Director — University of Colorado, Boulder; Douglas R Seals, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Clinical Translational Research Center, Boulder, Colorado, United States

REFERENCES:
- [Derived] Rossman MJ, Gioscia-Ryan RA, Santos-Parker JR, Ziemba BP, Lubieniecki KL, Johnson LC, Poliektov NE, Bispham NZ, Woodward KA, Nagy EE, Bryan NS, Reisz JA, D'Alessandro A, Chonchol M, Sindler AL, Seals DR. Inorganic Nitrite Supplementation Improves Endothelial Function With Aging: Translational Evidence for Suppression of Mitochondria-Derived Oxidative Stress. Hypertension. 2021 Apr;77(4):1212-1222. doi: 10.1161/HYPERTENSIONAHA.120.16175. Epub 2021 Mar 1. PMID 33641356
- [Derived] Jones AM, Vanhatalo A, Seals DR, Rossman MJ, Piknova B, Jonvik KL. Dietary Nitrate and Nitric Oxide Metabolism: Mouth, Circulation, Skeletal Muscle, and Exercise Performance. Med Sci Sports Exerc. 2021 Feb 1;53(2):280-294. doi: 10.1249/MSS.0000000000002470. PMID 32735111
- See also: description of our laboratory — https://www.colorado.edu/intphys/research/cardiovascular.html